CLINICAL TRIAL: NCT06667076
Title: A Phase 2b, Open-Label, Two-cohort Study of Subcutaneous Amivantamab in Combination With Lazertinib as First-Line Treatment, or Subcutaneous Amivantamab in Combination With Platinum-Based Chemotherapy as Second-line Treatment, for Common EGFR-Mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Amivantamab in Combination With Lazertinib, or Amivantamab in Combination With Platinum-Based Chemotherapy, for Common Epidermal Growth Factor Receptor (EGFR)-Mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Acronym: COPERNICUS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61186372NSC2012; 61186372NSC2012 (Other: Janssen Research & Development, LLC); 2025-520730-28-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab; lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Amivantamab and Lazertinib (Experimental): Participants will receive Amivantamab in combination with Lazertinib orally in 28-day cycles until disease progression, withdrawal of consent, death, or the investigator decides to discontinue treatment, whichever comes first.
  Interventions: Drug: Amivantamab; Drug: Lazertinib
- Cohort 2: Amivantamab and Chemotherapy (Experimental): Participants will receive Amivantamab in combination with chemotherapy (carboplatin and pemetrexed) intravenous (IV) infusion in 21-day cycles until disease progression, withdrawal of consent, death, or the investigator decides to discontinue treatment, whichever comes first.
  Interventions: Drug: Amivantamab; Drug: Chemotherapy: Pemetrexed; Drug: Chemotherapy: Carboplatin

INTERVENTIONS:
Drug: Amivantamab — Amivantamab will be administered.
  Other Names: JNJ-61186372
Drug: Lazertinib — Lazertinib tablet will be administered.
  Other Names: JNJ-73841937
  Arms: Cohort 1: Amivantamab and Lazertinib
Drug: Chemotherapy: Pemetrexed — Pemetrexed will be administered.
  Arms: Cohort 2: Amivantamab and Chemotherapy
Drug: Chemotherapy: Carboplatin — Carboplatin will be administered.
  Arms: Cohort 2: Amivantamab and Chemotherapy

SUMMARY:
The primary purpose of the study is to assess how well amivantamab in combination with lazertinib or in combination with chemotherapy works (antitumor activity) in participants with epidermal growth factor receptor mutated (EGFRm) non-small cell lung cancer (NSCLC; that is one of the major types of lung cancer).

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed advanced or metastatic non-small cell lung cancer (NSCLC) that is not amenable to curative intent therapy
* Epidermal growth factor resistance-mutation (EGFRm) must be an Ex19del or Ex21 L858R substitution, as detected by food and drug administration (FDA)-approved or other validated test in a clinical laboratory improvement amendments (CLIA)-certified laboratory (sites in the US), or an accredited local laboratory (sites outside of the US) in accordance with site standard of care. In the European union (EU), the local test must be Conformité Européenne (CE)-marked or an in-house laboratory-developed test from health institutions in the EU in accordance with Article 5(5) of the in vitro diagnostic regulations (IVDR ) 2071/746, as amended
* Have at least 1 measurable lesion, according to RECIST version (v)1.1, that has not been previously irradiated
* Any toxicities from prior systemic anticancer therapy must have resolved to national cancer institute common terminology criteria for adverse events (NCI-CTCAE) version 5.0 grade 1 or baseline level (except for alopecia [any grade], grade <=2 peripheral neuropathy, or grade <=2 hypothyroidism stable on hormone replacement)
* Have an eastern cooperative oncology group (ECOG) performance status of 0 to 1

Exclusion Criteria:

* Medical history of active interstitial lung disease (ILD), including drug-induced ILD or radiation pneumonitis. Participants with medical history of radiation pneumonitis, including radiation pneumonitis which required steroid treatment, should consult with the medical monitor and eligibility be assessed on a case-by-case basis
* Had major surgery excluding placement of vascular access or tumor biopsy or had significant traumatic injury within 4 weeks before the first dose of anticancer treatments or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study
* Participant has uncontrolled tumor-related pain (symptomatic lesions amenable to palliative radiotherapy should be treated prior to first dosing)
* Received an investigational treatment that has not been cleared (based on at least 5 half lives of any pharmaceutical treatment) before the planned first dose of study treatment or is currently enrolled in an investigational study
* Has a prior or concurrent second malignancy (other than the disease under study) which natural history or treatment could likely interfere with any study endpoints of safety or the efficacy of the study treatment(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2029-05-23 (Estimated); Study Completion 2030-12-26 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 4 Years and 6 months
  PFS is defined as the time from the date of first dose of any study treatment until the date of objective disease progression or death, whichever occurs first according to response evaluation criteria in solid tumors (RECIST) version (v) 1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
Number of Participants Reporting Dose Reductions, Interruptions, and Discontinuations | Up to 4 Years and 6 months
  Participants with dose reductions, interruptions, and discontinuations will be reported.
Number of Participants With Venous Thromboembolic Events (VTEs) | Up to 4 Years and 6 months
  Participants with signs and symptoms (dyspnea, tachypnea, upper- or lower-extremity swelling and discoloration) of VTE events, specifically pulmonary embolism, and deep vein thrombosis will be reported as monitored by the investigators.
Number of Participants With Dermatologic Adverse Events (AEs) | Up to 4 Years and 6 months
  Participants with dermatologic AEs will be reported.
Number of Participants with AEs by Severity | Up to 4 Years and 6 months
  Severity of AEs will be graded according to the national cancer institute common terminology criteria for adverse event (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening and Grade 5: death related to adverse event.
Overall Survival (OS) | Up to 4 Years and 6 months
  OS is defined as the time from the date of first dose of any study treatment until the date of death due to any cause.
Overall Response Rate (ORR) | Up to 4 Years and 6 months
  ORR is defined as the percentage of participants who achieve either a partial response (PR) or complete response (CR) as their best response both confirmed and unconfirmed, as defined using RECIST v1.1.
Clinical Benefit Rate (CBR) | Up to 4 Years and 6 months
  CBR is defined as the percentage of participants achieving CR or PR, both confirmed and unconfirmed, or durable stable disease (SD) of a duration of at least 11 weeks as defined using RECIST v1.1.
Duration of Response (DOR) | Up to 4 Years and 6 months
  DOR is defined as the time from the date of first documented response (PR or CR) until the date of documented progression or death, whichever occurs first, for participants who have PR or CR.
Time to Treatment Discontinuation (TTTD) | Up to 4 Years and 6 months
  TTTD is defined as the date from the date of first dose of any study treatment until discontinuation of study treatment for any reason, including disease progression, treatment toxicity or death, based on RECIST v 1.1.
Time to Subsequent Therapy (TTST) | Up to 4 Years and 6 months
  TTST is defined as the time from the date of first dose of any study treatment until the start date of the subsequent anticancer therapy following study treatment discontinuation or death, whichever occurs first.
Time to Symptomatic Progression (TTSP) | Up to 4 Years and 6 months
  TTSP is defined as the time from date of first dose of any study treatment to documentation in the electronic case report form (eCRF) of any of the following (whichever occurs earlier): onset of new symptoms or symptom worsening that is considered by the investigator to be related to lung cancer and requires either a change in systemic anticancer treatment and/or clinical intervention to manage symptoms or death.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (178):
- United States (147):
  - Southern Cancer Center, PC, Daphne, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - City of Hope Phoenix, Goodyear, Arizona
  - The Oncology Institute of Hope and Innovation, Cerritos, California
  - City of Hope Corona, Corona, California
  - City of Hope, Duarte, California
  - Providence Medical Foundation, Fullerton, California
  - Oncology Physicians Network Healthcare, Glendale, California
  - Los Angeles Cancer Network, Glendale, California
  - Glendale Adventist Medical Center, Glendale, California
  - Marin Cancer Center, Greenbrae, California
  - City of Hope Seacliff, Huntington Beach, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - University of California San Diego Health, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope Long Beach Elm, Long Beach, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Valkyrie Clinical Trials, Murrieta, California
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - St. Joseph Hospital Center for Cancer Prevention and Treatment, Orange, California
  - University of California Irvine, Orange, California
  - Sutter Health Palo Alto Medical Foundation, Palo Alto, California
  - Kaiser Permanente Roseville Medical Center, Roseville, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Sutter Institute for Medical Research, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - Kaiser Permanente San Francisco Medical Center, San Francisco, California
  - UCSF Zuckerberg San Francisco General Hospital, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Kaiser Permanente Santa Clara Medical Center, Santa Clara, California
  - Providence Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Northern California, Vallejo, California
  - Kaiser Permanente Walnut Creek Medical Center, Walnut Creek, California
  - John Muir Health Clinical Research Center, Walnut Creek, California
  - National Jewish Health, Denver, Colorado
  - Saint Josephs Hospital Cancer Centers of Colorado, Denver, Colorado
  - Lutheran Hospital Cancer Centers of Colorado, Golden, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Yale New Haven Hospital Yale Cancer Center, New Haven, Connecticut
  - ChristianaCare Helen F Graham Cancer Center and Research Institute, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - Baptist Lynn Cancer Institute, Boca Raton, Florida
  - The Oncology Institute of Hope and Innovation, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Univ of Florida, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Baptist Health Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists & Research Institute, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists & Research Institute, West Palm Beach, Florida
  - University Cancer And Blood Center LLC, Athens, Georgia
  - Grady Health System Correll Pavilion, Atlanta, Georgia
  - Piedmont Healthcare, Atlanta, Georgia
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - City of Hope Cancer Center, Newnan, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Illinois CancerCare, Peoria, Illinois
  - City of Hope Chicago, Zion, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Investigative Clinical Research of Indiana, LLC, Noblesville, Indiana
  - Accellacare of McFarland, Ames, Iowa
  - University of Kansas Cancer Center, Fairway, Kansas
  - University of Maryland, Baltimore, Maryland
  - Maryland Oncology Hematology P A, Silver Spring, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Trinity Health St Joseph Mercy Ann Arbor, Ypsilanti, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Jackson Oncology Associates, Jackson, Mississippi
  - Truman Medical Ctr West, Kansas City, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Hematology-Oncology Associates of CNY, East Syracuse, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - NYU Langone Health Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center Columbia University Medical Center, New York, New York
  - Ellis Hospital, Schenectady, New York
  - New York Cancer and Blood Specialists, Shirley, New York
  - Montefiore Medical Center, The Bronx, New York
  - Clinical Research Alliance Inc, Westbury, New York
  - Atrium Health, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Regional Medical Oncology Center, Wilson, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati Veterans Affairs Medical Center, Cincinnati, Ohio
  - Oncology Associates of Oregon PC Willamette Valley Cancer Institute, Eugene, Oregon
  - Oregon Health And Science University, Portland, Oregon
  - Lankenau Institute for Medical Research Main Line Health Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Lankenau Institute for Medical Research Main Line Health Paoli Hospital, Paoli, Pennsylvania
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Health Northeast, Philadelphia, Pennsylvania
  - McGlinn Cancer Institute Reading Hospital, West Reading, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Medical Group, Sioux Falls, South Dakota
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - University of Tennessee, Knoxville, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology South, Austin, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - Texas Oncology DFW, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Renovatio Clinical, El Paso, Texas
  - JPS Health Network, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Oncology Consultants Texas, Houston, Texas
  - Community Clinical Trials, Kingwood, Texas
  - Texas Oncology Odessa-West Texas Cancer Center, Odessa, Texas
  - Texas Oncology San Antonio Northeast, San Antonio, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - Texas Oncology - Northeast, Tyler, Texas
  - Texas Oncology-Gulf Coast, Webster, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Vista Oncology, Olympia, Washington
  - Summit Cancer Centers, Spokane, Washington
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Turku University Hospital, Turku
- France (3):
  - CHU de Brest - Hopital de la Cavale Blanche, Brest
  - CHU de Grenoble, La Tronche
  - I.C.O. Rene Gauducheau, Saint-Herblain
- St. Elisabeth Hospital Leipzig, Leipzig, Germany
- Greece (5):
  - Henry Dunant Hospital Center, Athens
  - Thoracic General Hospital Of Athens I Sotiria, Athens
  - Metaxa Cancer Center Hospital Of Piraeus, Piraeus
  - Anticancer Hospital of Thessaloniki Theageneio, Thessaloniki
  - Athens Medical Center S A Interbalkan Medical Center of Thessaloniki, Thessaloniki
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Ramat Gan
- Ospedale S. Maria Delle Croci, Ravenna, Italy
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Portugal (5):
  - Uls Braga - Hosp. Braga, Braga
  - Uls Alto Ave - Hosp. Sra. Da Oliveira Guimaraes, Braga
  - Hosp. Cuf Tejo, Lisbon
  - Uls Loures Odivelas - Hosp. Loures, Loures
  - Ipo Porto, Porto
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- Spain (3):
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
- United Kingdom (3):
  - Royal Marsden Hospital, London
  - Royal Marsden Hospital, Sutton
  - Torbay Hospital-Devon, Torquay

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency